CLINICAL TRIAL: NCT01734486
Title: Growth Response in Girls With Turner Syndrome During a Three-year GH Treatment Comparing Two Dose Regimens. Identification of Predictive Factors of Growth Response
Brief Title: Growth Response in Girls With Turner Syndrome
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GHTUR/F/3
Record Dates: First submitted 2012-11-22; First posted 2012-11-27 (Estimated); Last update posted 2017-02-28 (Actual); Status verified 2017-02

CONDITIONS: Genetic Disorder; Turner Syndrome
MeSH Terms: conditions — Genetic Diseases, Inborn; Turner Syndrome | interventions — Human Growth Hormone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Low dose (Experimental)
  Interventions: Drug: somatropin
- High dose (Experimental)
  Interventions: Drug: somatropin

INTERVENTIONS:
Drug: somatropin — 0.9 UI/kg/week. Subcutaneous injection for 3 years
  Arms: Low dose
Drug: somatropin — 1.8 UI/kg/week. Subcutaneous injection for 3 years
  Arms: High dose

SUMMARY:
This trial is conducted in Europe. The aim of the trial is to evaluate growth response of two somatropin dose regimens in girls with Turner Syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Turner syndrome
* If age below 3 years, either body height below - 1 SD (standard deviation) with average growth velocity according to chronological age or body height below 0 SD with growth velocity below -1 SD according to chronological age
* If age above 3 years, body height below - 1 SD with average growth velocity according to chronological age
* Measured parental height available
* Written informed consent

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 1996-09-23 (Actual); Primary Completion 2003-05-21 (Actual); Study Completion 2003-05-21 (Actual)

PRIMARY OUTCOMES:
Height gain, SDS (Standard Deviation Score)
Height gain in cm

SECONDARY OUTCOMES:
Height
Bone maturation

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (15):
- France (15):
  - Novo Nordisk Investigational Site, Besançon
  - Novo Nordisk Investigational Site, Bordeaux
  - Novo Nordisk Investigational Site, Dunkirk
  - Novo Nordisk Investigational Site, Grenoble
  - Novo Nordisk Investigational Site, Lille
  - Novo Nordisk Investigational Site, Lorient
  - Novo Nordisk Investigational Site, Nice
  - Novo Nordisk Investigational Site, Paris
  - Novo Nordisk Investigational Site, Reims
  - Novo Nordisk Investigational Site, Rennes
  - Novo Nordisk Investigational Site, Rouen
  - Novo Nordisk Investigational Site, Tarbes
  - Novo Nordisk Investigational Site, Toulouse
  - Novo Nordisk Investigational Site, Tours
  - Novo Nordisk Investigational Site, Vandœuvre-lès-Nancy

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com